CLINICAL TRIAL: NCT00145314
Title: 5-Fluorouracil/Folinate/Oxaliplatin (Eloxatin) (FLOX Regimen), Given Continuously or Intermittently, in Combination With Cetuximab (Erbitux), in First-line Treatment of Metastatic Colorectal Cancer. A Phase III Multicenter Trial.
Brief Title: FLOX in Combination With Cetuximab in First-line Treatment of Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Nordic Colorectal Cancer Biomodulation Group (Other)
Responsible Party: Kjell M. Tveit, MD, PhD, The Nordic Colorectal Cancer Biomodulation Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nordic VII; EudraCT no.: 2005-000117-34
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; FLOX; Cetuximab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Cetuximab; Leucovorin; Oxaliplatin

ARMS (3):
- A (Active Comparator): FLOX: 5-fluorouracil/folinic acid/oxaliplatin; Nordic Regimen; given continuosly
  Interventions: Drug: FLOX (5-fluorouracil/folinic acid/oxaliplatin)
- B (Experimental): FLOX: 5-fluorouracil/folinic acid/oxaliplatin and cetuximab
  Interventions: Drug: FLOX (5-fluorouracil/folinic acid/oxaliplatin) and Cetuximab
- C (Experimental): FLOX given intermittently and maintenance cetuximab
  Interventions: Drug: FLOX (5-fluorouracil and folinic acid and oxaliplatin) intermittently and maintenance cetuximab

INTERVENTIONS:
Drug: FLOX (5-fluorouracil/folinic acid/oxaliplatin) — FLOX every 2nd week
  Arms: A
Drug: FLOX (5-fluorouracil/folinic acid/oxaliplatin) and Cetuximab — FLOX every 2nd week Cetuximab weekly
  Arms: B
Drug: FLOX (5-fluorouracil and folinic acid and oxaliplatin) intermittently and maintenance cetuximab — FLOX every 2nd week for 8 cycles. Stop of FLOX until progression then FLOX is reintroduced.
  Cetuximab weekly.
  Arms: C

SUMMARY:
The main objective of this trial is to explore the effect of combining an established chemotherapy regimen (FLOX), based on 5-fluorouracil, folinic acid, and oxaliplatin (Eloxatin®), with the EGF receptor antibody cetuximab (Erbitux®) in first-line treatment of metastatic colorectal cancer. The trial will investigate two regimens of FLOX plus cetuximab, in which FLOX is given continuously or intermittently, compared to standard FLOX without cetuximab.

ELIGIBILITY:
Inclusion Criteria:

Histology and staging disease:

* Histological proven adenocarcinoma of the colon or rectum;
* At least one measurable metastatic disease
* If only one metastatic lesion and no S-CEA elevation, histology is mandatory;
* Availability of tumour sample for EGFR assessment.

General conditions:

* Age >18 and < 75 years;
* WHO performance status: life expectancy of more than 3 months;
* Adequate haematological function
* Adequate renal and hepatic functions
* Written informed consent

Exclusion Criteria:

Prior therapy:

* No prior chemotherapy for advanced/metastatic disease;
* No adjuvant chemotherapy the last 6 months before inclusion;
* No previous oxaliplatin;

Prior or current history:

* No current indication for resection with a curative intent;
* No evidence of CNS metastasis;
* No current infection, unresolved bowel obstruction or subobstruction, uncontrolled Crohn's disease or ulcerative colitis;
* No current history of chronic diarrhoea;
* No peripheral neuropathy;
* No other serious illness or medical conditions (including contraindication to 5 FU e.g.: angor, myocardial infarction within 6 months, contraindications to monoclonal antibodies);
* No past or concurrent history of malignant neoplasm other than colorectal adenocarcinoma within the past five years, except curatively treated non melanoma skin cancer or in situ carcinoma of the cervix;

Concomitant treatments:

* No concomitant (or within 4 weeks before randomisation) administration of any other experimental drug under investigation;
* No concurrent treatment with any other anti-cancer therapy;

Other:

* Not pregnant, no breast feeding
* Fertile patients must use adequate contraceptives
* Not include patients clearly intending to withdraw from the study if not randomised in the willing arm or patients who cannot be regularly followed up for psychological, social, familiar or geographic reasons.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2005-05; Primary Completion 2009-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To compare efficacy, as measured by time to disease progression, of treatment with cetuximab in combination with the FLOX regimen compared to FLOX alone, in first- line treatment of patients with metastatic cororectal cancer | Every 4th cycle

SECONDARY OUTCOMES:
To measure response rates, response duration, secondary surgical curative resection frequency, safety profile, overall survival and quality of life in the treatment groups. | Every 2nd week (safety profile)

CONTACTS AND LOCATIONS:
Overall Officials: Kjell M. Tveit, MD, PhD, Principal Investigator — Professor at Ullevål University Hospital, Norway
Locations (1):
- The Nordic Colorectal Cancer Biomodulation Group, Oslo, Norway

REFERENCES:
- [Derived] Hamfjord J, Guren TK, Glimelius B, Sorbye H, Pfeiffer P, Dajani O, Lingjaerde OC, Tveit KM, Spindler KG, Pallisgaard N, Kure EH. Exploring Early Kinetic Profiles of CEA, ctDNA and cfDNA in Patients With RAS-/BRAF-Mutated Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2025 Jun;24(2):153-158. doi: 10.1016/j.clcc.2024.11.004. Epub 2024 Dec 3. PMID 39743478
- [Derived] Hamfjord J, Guren TK, Dajani O, Johansen JS, Glimelius B, Sorbye H, Pfeiffer P, Lingjaerde OC, Tveit KM, Kure EH, Pallisgaard N, Spindler KG. Total circulating cell-free DNA as a prognostic biomarker in metastatic colorectal cancer before first-line oxaliplatin-based chemotherapy. Ann Oncol. 2019 Jul 1;30(7):1088-1095. doi: 10.1093/annonc/mdz139. PMID 31046124
- [Derived] Kjersem JB, Thomsen M, Guren T, Hamfjord J, Carlsson G, Gustavsson B, Ikdahl T, Indrebo G, Pfeiffer P, Lingjaerde O, Tveit KM, Wettergren Y, Kure EH. AGXT and ERCC2 polymorphisms are associated with clinical outcome in metastatic colorectal cancer patients treated with 5-FU/oxaliplatin. Pharmacogenomics J. 2016 Jun;16(3):272-9. doi: 10.1038/tpj.2015.54. Epub 2015 Aug 11. PMID 26261061
- [Derived] Kjersem JB, Skovlund E, Ikdahl T, Guren T, Kersten C, Dalsgaard AM, Yilmaz MK, Fokstuen T, Tveit KM, Kure EH. FCGR2A and FCGR3A polymorphisms and clinical outcome in metastatic colorectal cancer patients treated with first-line 5-fluorouracil/folinic acid and oxaliplatin +/- cetuximab. BMC Cancer. 2014 May 19;14:340. doi: 10.1186/1471-2407-14-340. PMID 24884501
- [Derived] Kjersem JB, Ikdahl T, Guren T, Skovlund E, Sorbye H, Hamfjord J, Pfeiffer P, Glimelius B, Kersten C, Solvang H, Tveit KM, Kure EH. Let-7 miRNA-binding site polymorphism in the KRAS 3'UTR; colorectal cancer screening population prevalence and influence on clinical outcome in patients with metastatic colorectal cancer treated with 5-fluorouracil and oxaliplatin +/- cetuximab. BMC Cancer. 2012 Nov 20;12:534. doi: 10.1186/1471-2407-12-534. PMID 23167843